CLINICAL TRIAL: NCT07396675
Title: Improving Postoperative Debriefings: the Added Value of Operating Room Black Box Supported Debriefings and Their Effect on Healthcare Professionals Perceived Effectiveness and Psychological Safety.
Brief Title: Operating Room Black Box Supported Debriefings and Their Effect on Healthcare Professionals Effectiveness and Psychological Safety.
Acronym: ORBLACKBOX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ORNND - Operating Room Nurse Network Denmark (Network)
Collaborators: Rigshospitalet, Denmark (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Johanne Søborg Hartmann, Principal investigator, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KEEPCARING EU Debriefing WP3
Record Dates: First submitted 2025-08-14; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-08

CONDITIONS: Stress; Resilience; Psychological Safety; Burnout, Healthcare Workers; Teamwork
Keywords: debriefing; teamwork; psychological safety; operating room; operating room black box
MeSH Terms: conditions — Burnout, Psychological | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Debriefings with Operating Room Black Box audio and video material (Other): Operating Room Black Box audio and video material included in debriefings
  Interventions: Behavioral: Debriefing
- Debriefings without Operating Room Black Box audio and video material (Other): Debriefings without Operating Room Black Box audio and video material
  Interventions: Behavioral: Debriefing
- Observation of team debriefing (Other): Observational study part of team member interaction during the team debriefing
  Interventions: Behavioral: Debriefing
- Qualitative interviews after team debriefing (Other): Qualitative interview study part of team members after debriefing
  Interventions: Behavioral: Debriefing

INTERVENTIONS:
Behavioral: Debriefing — Debriefing after surgery for operating room staff

SUMMARY:
This study is enrolled in the European KEEPCARING Project. KEEPCARING aims to (re-)build wellbeing and resilience of healthcare workforce in EU hospitals by co-creating a multi-faceted non-digital, digital, and AI-supported solution package to prevent burnout among (aspirant) healthcare professionals on the individual, team, and organizational level.

This study specifically investigate the operating room staff wellbeing and resilience. The healthcare system is currently struggling to retain and attract operating room personnel. A factor of importance to consider here is occupational stress. If not recognized or mitigated well, occupational stress and personal efficacy can eventually evolve into a syndrome labelled as 'burnout'. In addition, communication and resilience patterns between operating room staff members are of influence, poor and/or inadequate communication among staff may be a factor of stress, compromising their work and wellbeing. In contrast, communication patterns that have a high standard and clarity may support resilience. The ability to speak up and being able to advocate concerns of all team members is of the highest importance here. Indeed, psychological safety and effective teamwork patterns are key for the working environment, performance, patient safety, and job satisfaction. To prevent mistakes during surgery, a safe space where team members can freely speak up is vital.

To improve psychological safety, and teamwork among OR staff, team debriefing after surgery is known to be effective. What is not known; is whether team debriefing with the additional support derived from audio- and video recordings of the surgery is equally effective as debriefing without.

The objective of this study is to evaluate the impact of structured postoperative debriefings with and without procedural, structured audio- and video recordings, on team performance, psychological safety, and non-technical skills in the operating room. Specifically, this study aims to compare augmented debriefings with non-augmented debriefings, to assess differences in perceived usefulness, psychological safety, and observed improvements in teams' non-technical skills.

This is an international quasi-experimental comparative study. The intervention consists of postoperative team debriefing using audio and video recordings ('augmented debriefing') from Operating Room Black Box system provided by Surgical Safety Technologies. The control group will have a postoperative team debriefing that is not augmented with Operating Room Black Box derived data. An identical debriefing template will be designed for both groups.

DETAILED DESCRIPTION:
Design and setting This is an international quasi-experimental comparative study, following the guidelines for complex interventions in health. The intervention will be ORBB augmented team-debriefing after surgery. The control group will debrief after surgery without the assistance of the ORBB. An identical debriefing template has been designed for both groups.

This study will be conducted at OR departments in three university hospitals, located in three different countries: Rigshospitalet, Copenhagen University Hospital (RIGS), Amsterdam University Medical Center (AUMC) and University Medical Center Hamburg-Eppendorf (UKE). RIGS have nine OR's with ORBB installed and access to ORBB-generated video material and outcome reports using explainable AI. AUMC is expected to have two OR's with ORBB installed before beginning of study. RIGS and AUMC are planned as both interventions and control sites, AUMC will if unforeseen delays occur with ORBB installation, be a control site (e.g. have only non-augmented debriefings). UKE does not have ORBB and will be a control site.

Characteristics of the study population

Participants Full OR teams performing elective daytime surgeries, approximately 4-12 people per team. The teams will be selected from a variety of specialties such as cardiothoracic, gynecology, urology, abdominal, vascular, and orthopedic surgery. Depending on the variety and possibility at each site, RIGS, AUMC and UKE, including limitations due to which ORs have ORBB installed.

Intervention Investigators anticipate that the intervention of the study occurs over a 1-month period for each team. In total, the intervention period is scheduled over a one-year period within 2026. During all data collection team members speak in their native language, so for RIGS this is Danish, for AUMC Dutch and for UKE German. The intervention includes a baseline questionnaire, a surgery, a short questionnaire after surgery, an observed debriefing and a follow up questionnaire after surgery.

The intervention set up is the same for teams with and without ORBB, only difference is the audio and video from the ORBB and SST. Furthermore, the debriefings will be audio recorded, and a researcher will observe the sessions. After the intervention period, a sample of participants will be asked to participate in a qualitive interview study.

Preparation before team debriefing After surgery the OR team members individually fill out a short questionnaire. Team members will answer questions about the following four topics: overall procedure, teamwork, safety protocols and learning opportunities.

The key points are wide in their definitions purposely because the team members should have the possibility to choose meaningful moments from the actual OR situation within the four topics. They must answer the questionnaire within 12 hours after surgery, to secure that the OR episode is still fresh in their minds.

Afterwards the researcher on site will review the questionnaires and during non-augmented debriefings bring their answers into play. During augmented debriefings, the researcher will 'flag' the surgery within the SST platform and in collaboration with SST create 3-4 videoclips, that contains the key elements chosen by the team members.

Team debriefing The setup in both augmented and non-augmented debriefings focus on creating a dedicated learning environment that prioritizes reflection, open communication, and psychological safety during the sessions. The physical space is carefully designed to support these critical aspects of team learning and collaboration.

In every debriefing an independent educational specialist (with no formal or working relation to the OR) is used as a moderator that controls the conversation and follow the debriefing template.

During the debriefing a researcher observes the conversation and interactions between team members and the moderator. The observing researcher sits in a corner of the room, disturbing as little as possible, being quiet and only taking field notes of the interaction between the team members and the moderator. The debriefing sessions will be audio-recorded, and transcribed verbatim by the observing researcher.

The session is time-limited to 30-60 minutes, balancing comprehensive discussion with efficiency. Critically, the debriefing is ideally conducted after approximately 5 (to a maximum of 15 days) following the surgery, allowing team members sufficient time to process the experience while maintaining the immediacy of relevant insights and reflections emotionally and professionally.

At the same time, securing the researchers a timespan to overview the short questionnaires, and select key points, for the moderator to work with in the debriefing sessions. Specific for the ORBB augmented debriefings, at the same time securing a timespan for the researchers to select and prepare 3-4 videoclips within the ORBB platform in collaboration with SST before the debriefing.

Debriefing template for debriefing In this study investigators implement a six-step team debriefing model, tested with a high rate of participant satisfaction (7.8/10 rating) in a previous study on 35 ORBB augmented abdominal surgery team debriefing sessions. The researchers concluded that their proposed approach effectively facilitates OR debriefing across diverse healthcare settings and provides a viable framework for establishing a much-needed debriefing culture to enhance surgical team performance. Investigators adjusted the model with few moderations to fit both OR debriefings with and without ORBB augmented data, and to include more OR specialties, on top of abdominal OR teams.

During the debriefings the moderator controls the conversation, and every team member represents their field of expertise in the OR. The moderator follows the themes; experience, observation, analyze and application.

During the debriefings all teams will focus on psychological safety and problem solving within the following four key points: overall procedure, teamwork, safety protocols and learning opportunities. For the intervention sites, the debriefing templates are the same as the control site, only add on is the ORBB augmented material of 3-4 videoclips and objective data from SST platform, integrated into the debriefing templates.

Data and Outcomes Investigators will gather data about the debriefings and measure outcomes through the following measurement tools; observation and audio recording of team debriefings, individual pre- and post-debriefing questionnaires and qualitative interviews. Specifically for surgeries using the ORBB system, OR teams will also be observed through audio and video-review from ORBB, including AI statistical data provided by SST.

This will allow for in-depth analysis of team dynamics, providing a structured approach to understanding and improving collaborative practices in surgical settings. By capturing both quantitative ratings and qualitative insights, the research aims to develop targeted strategies that can elevate team communication, psychological safety, and overall performance.

Regulatory and ethics The coordinating hospital for this study is RIGS. In 2019, the Danish Data Protection Agency approved the overall ORBB project (registration no.: VD-2019-275). The project was submitted to the Regional Ethics Committee in 2018, and no ethical approval was needed (registration no.: H-18018801). Additional approval for this debriefing study has been obtained in 2025 from the Regional Legal and Ethics Committee in Copenhagen, Denmark, PRIVACY - legal GRC (ID-NUMBER: p-2025-19044).

Participation in this study is voluntary and thus consent based. All participants will receive oral and written information before entering the study, and they must sign a consent form to participate. Participants can withdraw their consent at any time. Informed consent forms will be automatically uploaded to certified servers of Castor. Data will be stored on certified servers of Zenodo, which complies with all regulations and applicable laws. Data will also be stored locally in the department's computer system drive.

ELIGIBILITY:
Inclusion Criteria:

* Participants work in an OR-team at RIGS, AUMC or UKE.
* Participants must have given informed written consent to participate in the study.
* Participants must be in the OR for the majority of the procedure or/and have a central role in the teamwork.
* At RIGS and AUMC participants for the ORBB debriefings must also be part of teams conducting surgeries in the OR where ORBB is installed (not all ORs have ORBB).
* Participants can either be surgeons, anesthesiologist, anesthesia nurses, residents, OR-nurses, perfusionists, interns, nurse students or other OR-staff.

Exclusion Criteria:

* Visitors, guests, and other staff only watching the surgery, are excluded from participation.
* Individuals who are unable or unwilling to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Psychological safety | 1-3 months
  Amy Edmondsons Scale on psychological safety and learning behaviour in operating room teams. 7 items scale; minimum value 1, maximum value 5.
Usefulness and satisfaction of the team-debriefing | 1-3 months
  Usefulness and satisfaction of the team-debriefing, Van Dalen scale. 6 items score, minimum value 1, maximum value 5.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] The ethnographic interview af James P. Spradley
- [Background] Brinkmann S, Kvale S. Interviews: Learning the craft of qualitative research interviewing. 3rd ed. Thousand Oaks: CA: Sage; 2003.
- [Background] Oakley A, Strange V, Bonell C, Allen E, Stephenson J. Process evaluation in randomised controlled trials of complex interventions. BMJ. 2006 Feb 18;332(7538):413-6.
- [Background] Rose Gillian. Visual methodologies : an introduction to researching with visual materials. 2023;454.
- [Background] Cook DA, Brydges R, Ginsburg S, Hatala R. A contemporary approach to validity arguments: A practical guide to Kane's framework. Med Educ. 2015 Jun 1;49(6):560-75.
- [Background] Spradley JP. Qualitative Research Guide: Participant Observation. Holt, Rinehart and Winston, Inc
- [Background] Yule S, Flin R, Paterson-Brown S, Maran N, Rowley D. Development of a rating system for surgeons' non-technical skills. Med Educ. 2006 Nov;40(11):1098-104. doi: 10.1111/j.1365-2929.2006.02610.x. PMID 17054619
- [Background] Gaba DM. Crisis resource management and teamwork training in anaesthesia. Br J Anaesth. 2010 Jul;105(1):3-6. doi: 10.1093/bja/aeq124. No abstract available. PMID 20551023
- [Background] Biesta GJJ, van Braak M. Beyond the Medical Model: Thinking Differently about Medical Education and Medical Education Research. Teach Learn Med. 2020 Aug 7;32(4):449-56.
- [Background] Gadamer HG. Truth and method. Bloomsbury Academic; 1960.
- [Background] Cantor GN, Bhaskar R. The Possibility of Naturalism: A Philosophical Critique of the Contemporary Human Sciences. Philos Q. 1982 Jul;32(128):280.
- [Background] Alvesson Mats, Sköldberg Kaj. Reflexive methodology : new vistas for qualitative research. 2018;437.
- [Background] Cheng A, Eppich W, Grant V, Sherbino J, Zendejas B, Cook DA. Debriefing for technology-enhanced simulation: a systematic review and meta-analysis. Med Educ. 2014 Jul;48(7):657-66. doi: 10.1111/medu.12432. PMID 24909527
- [Background] Nembhard IM, Edmondson AC. Making it safe: The effects of leader inclusiveness and professional status on psychological safety and improvement efforts in health care teams. J Organ Behav
- [Background] Hallberg Ingalill, Richards DA. Complex interventions in health : an overview of research methods
- [Background] Shanafelt TD, Balch CM, Bechamps G, Russell T, Dyrbye L, Satele D, et al. Burnout and Medical Errors Among American Surgeons. Ann Surg. 2010 Jun;251(6):995-1000.
- [Background] Langerman A, Grantcharov TP. Are We Ready for Our Close-up?: Why and How We Must Embrace Video in the OR. Ann Surg. 2017 Dec;266(6):934-936. doi: 10.1097/SLA.0000000000002232. No abstract available. PMID 28338514
- [Background] Møller EK, Sørensen JL, Topperzer MK, Koerner C, Ottesen B, Rosendahl M, et al. Implementation of an innovative technology called the OR Black Box: A feasibility study. Surgical Innovation SAGE. 2023;30(1):64-72.
- [Background] Rose MR, Rose KM. Use of a Surgical Debriefing Checklist to Achieve Higher Value Health Care. Am J Med Qual. 2018 Sep/Oct;33(5):514-522. doi: 10.1177/1062860618763534. Epub 2018 Apr 2. PMID 29606010
- [Background] Leonard LD, Shaw M, Moyer A, Tevis S, Schulick R, McIntyre R Jr, Ballou M, Reiter K, Lace C, Weitzel N, Wiler J, Meacham R, Cumbler E, Steward L. The surgical debrief: Just another checklist or an instrument to drive cultural change? Am J Surg. 2022 Jan;223(1):120-125. doi: 10.1016/j.amjsurg.2021.07.043. Epub 2021 Jul 29. PMID 34407917
- [Background] Mundt AS, Gjeraa K, Spanager L, Petersen SS, Dieckmann P, Ostergaard D. Okay, let's talk - short debriefings in the operating room. Heliyon. 2020 Jul 4;6(7):e04386. doi: 10.1016/j.heliyon.2020.e04386. eCollection 2020 Jul. PMID 32671270
- [Background] Skegg E, McElroy C, Mudgway M, Hamill J. Debriefing to improve interprofessional teamwork in the operating room: A systematic review. J Nurs Scholarsh. 2023 Nov;55(6):1179-1188. doi: 10.1111/jnu.12924. Epub 2023 Jul 15. PMID 37452720
- [Background] McElroy C, Skegg E, Mudgway M, Murray N, Holmes L, Weller J, et al. Psychological Safety and Hierarchy in Operating Room Debriefing: Reflexive Thematic Analysis. Journal of Surgical Research. 2024 Mar 1;295:567-73.
- [Background] Boet S, Sharma B, Pigford AA, Hladkowicz E, Rittenhouse N, Grantcharov T. Debriefing decreases mental workload in surgical crisis: A randomized controlled trial. Surgery. 2017 May;161(5):1215-1220. doi: 10.1016/j.surg.2016.11.031. Epub 2017 Jan 16. PMID 28104293
- [Background] Wright MI, Polivka B, Abusalem S. An Examination of Factors That Predict the Perioperative Culture of Safety. AORN J. 2021 May 1;113(5):465-75.
- [Background] Weller JM, Long JA. Creating a climate for speaking up. Br J Anaesth. 2019 Jun 1;122(6):710-3.
- [Background] Maunder R et. al. Burnout in hospital-based healthcare workers during COVID-19. . Science Briefs of the Ontario COVID-19 Science Advisory Table. 2021;
- [Background] Al Abbas AI, Meier J, Daniel W, Cadeddu JA, Bartolome S, Willett DL, et al. Impact of team performance on the surgical safety checklist on patient outcomes: an operating room black box analysis. Surg Endosc
- [Background] Feo R, Kitson A. Promoting patient-centred fundamental care in acute healthcare systems. Int J Nurs Stud. 2016 May;57:1-11. doi: 10.1016/j.ijnurstu.2016.01.006. Epub 2016 Feb 1. PMID 27045560
- [Background] Arakelian E, Swenne CL, Lindberg S, Rudolfsson G, von Vogelsang AC. The meaning of person-centred care in the perioperative nursing context from the patient's perspective - an integrative review. J Clin Nurs. 2017 Sep;26(17-18):2527-2544. doi: 10.1111/jocn.13639. Epub 2017 Feb 16. PMID 27862496
- [Background] Balch CM, Shanafelt T. Combating Stress and Burnout in Surgical Practice: A Review. Adv Surg. 2010 Sep;44(1):29-47.
- [Background] Li N, Zhang L, Li X, Lu Q. The influence of operating room nurses' job stress on burnout and organizational commitment: The moderating effect of over-commitment. J Adv Nurs
- [Background] Tekeletsadik S, Mulat H, Necho M, Waja T. Occupational Stress and Its Associated Factors among Health Care Professionals Working At a Setting of a Specialized Mental Hospital, Addis Ababa, Ethiopia, 2017: A Hospital-Based Cross-Sectional Study. J Psychol Psychother
- [Background] Magnavita N, Soave PM, Ricciardi W, Antonelli M. Occupational Stress and Mental Health among Anesthetists during the COVID-19 Pandemic. Int J Environ Res Public Health. 2020 Nov 8;17(21):8245. doi: 10.3390/ijerph17218245. PMID 33171618
- [Background] Yosef B, Woldegerima Berhe Y, Yilkal Fentie D, Belete Getahun A. Occupational Stress among Operation Room Clinicians at Ethiopian University Hospitals. J Environ Public Health. 2022 Jan 19;2022(1).
- [Background] Aiken LH, Sloane DM, Bruyneel L, Van den Heede K, Griffiths P, Busse R, et al. Nurse staffing and education and hospital mortality in nine European countries: a retrospective observational study.
- [Background] Pattni N, Arzola C, Malavade A, Varmani S, Krimus L, Friedman Z. Challenging authority and speaking up in the operating room environment: a narrative synthesis. Br J Anaesth. 2019 Feb 1;122(2):233-44.
- [Background] Arad D, Finkelstein A, Rozenblum R, Magnezi R. Patient safety and staff psychological safety: A mixed methods study on aspects of teamwork in the operating room. Front Public Health. 2022 Dec 23;10.
- [Background] Mayes CG, Cochran K. Factors Influencing Perioperative Nurse Turnover: A Classic Grounded Theory Study. AORN J. 2023 Mar;117(3):161-174. doi: 10.1002/aorn.13880. PMID 36825918
- [Background] Birkbak A. Actor-Network Theory. Sociology
- [Background] Tørring B, Gittell JH, Laursen M, Rasmussen BS, Sørensen EE. Communication and relationship dynamics in surgical teams in the operating room: An ethnographic study. BMC Health Serv Res. 2019 Jul 29;19(1).
- [Background] Schaap M, Hanskamp-Sebregts M, Merkx T (M. AW), Heideveld-Chevalking A (A. J), Meijerink J (W. JHJ). Long-term effects of perioperative briefing and debriefing on team climate: A mixed-method evaluation study. Int J Clin Pract. 2021 Mar 21;75(3).
- [Background] Sandelin A, Kalman S, Gustafsson BA. Prerequisites for safe intraoperative nursing care and teamwork-Operating theatre nurses' perspectives: A qualitative interview study. J Clin Nurs. 2019 Jul;28(13-14):2635-2643. doi: 10.1111/jocn.14850. Epub 2019 Mar 29. PMID 30865340
- [Background] van Dalen ASHM, van Haperen M, Swinkels JA, Grantcharov TP, Schijven MP. Development of a Model for Video-Assisted Postoperative Team Debriefing. Journal of Surgical Research. 2021 Jan;257:625-35.
- [Background] Goldenberg MG, Jung JJ, Grantcharov T. Using data to enhance performance and improve quality and safety in surgery. JAMA Surg. 2017;152(10).
- [Background] Mitchell L, Flin R, Yule S, Mitchell J, Coutts K, Youngson G. Development of a behavioural marker system for scrub practitioners' non-technical skills (SPLINTS system). J Eval Clin Pract. 2013 Apr;19(2):317-23. doi: 10.1111/j.1365-2753.2012.01825.x. Epub 2012 Apr 15. PMID 22502593
- [Background] Fletcher G, Flin R, McGeorge P, Glavin R, Maran N, Patey R. Anaesthetists' Non-Technical Skills (ANTS): evaluation of a behavioural marker system † †Declaration of interest: The ANTS system was developed under research funding from the Scottish Council for Postgraduate Medical and Dental Education, now part of NHS Education for Scotland, through grants to the University of Aberdeen from September 1999 to August 2003. The views presented in this paper are those of the authors and should not be taken to represent the position or policy of the funding body. Br J Anaesth. 2003 May;90(5):580-8.
- [Background] Whittaker G, Abboudi H, Khan MS, Dasgupta P, Ahmed K. Teamwork Assessment Tools in Modern Surgical Practice: A Systematic Review. Surg Res Pract. 2015;2015:494827. doi: 10.1155/2015/494827. Epub 2015 Sep 3. PMID 26425732
- [Background] Zuckerman SL, France DJ, Green C, Leming-Lee S, Anders S, Mocco J. Surgical debriefing: a reliable roadmap to completing the patient safety cycle. Neurosurg Focus. 2012 Nov;33(5):E4. doi: 10.3171/2012.8.FOCUS12248. PMID 23116099
- [Background] Hamad GG, Brown MT, Clavijo-Alvarez JA. Postoperative video debriefing reduces technical errors in laparoscopic surgery. Am J Surg. 2007 Jul;194(1):110-4. doi: 10.1016/j.amjsurg.2006.10.027. PMID 17560921
- [Background] Jung JJ, Jüni P, Lebovic G, Grantcharov T. First-year analysis of the Operating Room Black Box. Ann Surg. 2018;
- [Background] van Dalen ASHM, Jansen M, van Haperen M, van Dieren S, Buskens CJ, Nieveen van Dijkum EJM, et al. Implementing structured team debriefing using a Black Box in the operating room: surveying team satisfaction. Surg Endosc. 2021 Mar 1;35(3):1406-19.
- [Background] Rudolph JW, Simon R, Raemer DB, Eppich WJ. Debriefing as formative assessment: closing performance gaps in medical education. Acad Emerg Med. 2008 Nov;15(11):1010-6. doi: 10.1111/j.1553-2712.2008.00248.x. Epub 2008 Oct 20. PMID 18945231
- [Background] Sawyer T, Eppich W, Brett-Fleegler M, Grant V, Cheng A. More Than One Way to Debrief. Simulation in Healthcare: The Journal of the Society for Simulation in Healthcare. 2016 Jun;11(3):209-17.
- [Background] McElroy C, Skegg E, Mudgway M, Murray N, Holmes L, Weller J, et al. Psychological Safety and Hierarchy in Operating Room Debriefing: Reflexive Thematic Analysis. Journal of Surgical Research. 2024 Mar;295:567-73.
- [Background] Fanning RM, Gaba DM. The Role of Debriefing in Simulation-Based Learning. Simulation in Healthcare: The Journal of the Society for Simulation in Healthcare. 2007;2(2):115-25.
- [Background] Leonard M. The human factor: the critical importance of effective teamwork and communication in providing safe care. Qual Saf Health Care. 2004 Oct 1;13(suppl_1):i85-90.
- [Background] Speaking Up in the Operating Room: How Team Leaders Promote Learning in Interdisciplinary Action Teams - Edmondson - 2003 - Journal of Management Studies - Wiley Online Library
- [Background] Edmondson A. Psychological safety and learning behavior in work teams. Adm Sci Q. 1999;44(2):350-83.
- [Background] Schonfeld IS, Bianchi R. Burnout and Depression: Two Entities or One? J Clin Psychol. 2016 Jan;72(1):22-37. doi: 10.1002/jclp.22229. Epub 2015 Oct 9. PMID 26451877
- [Background] Schaufeli WB, Desart S, De Witte H. Burnout Assessment Tool (BAT)-Development, Validity, and Reliability. Int J Environ Res Public Health. 2020 Dec 18;17(24):9495. doi: 10.3390/ijerph17249495. PMID 33352940
- [Background] Epel ES, Crosswell AD, Mayer SE, Prather AA, Slavich GM, Puterman E, et al. More than a feeling: A unified view of stress measurement for population science. Front Neuroendocrinol
- [Background] Bianchi R, Lindsäter E, Vollan TE, Tesaker R, Mathisen HH, Øyangen SH, et al. Most people do not attribute their burnout symptoms to work. J Psychosom Res
- [Background] Bianchi R, Schonfeld IS, Laurent E. The Trouble With Burnout: An Update on Burnout-Depression Overlap. Am J Psychiatry. 2019 Jan 1;176(1):79. doi: 10.1176/appi.ajp.2018.18091026. No abstract available. PMID 30848942
- [Background] Williams ES, Manwell LB, Konrad TR, Linzer M. The relationship of organizational culture, stress, satisfaction, and burnout with physician-reported error and suboptimal patient care: results from the MEMO study. Health Care Manage Rev. 2007 Jul-Sep;32(3):203-12. doi: 10.1097/01.HMR.0000281626.28363.59. PMID 17666991
- [Background] Edu-Valsania S, Laguia A, Moriano JA. Burnout: A Review of Theory and Measurement. Int J Environ Res Public Health. 2022 Feb 4;19(3):1780. doi: 10.3390/ijerph19031780. PMID 35162802
- [Background] McGonigal Kelly. The upside of stress : why stress is good for you, and how to get good at it. 2016 .
- [Background] Lu S, Wei F, Li G. The evolution of the concept of stress and the framework of the stress system. Cell Stress. 2021;5(6):76.
- [Background] Chu B, Marwaha K, Sanvictores T, Awosika AO, Ayers D. Physiology, Stress Reaction. 2024 May 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK541120/ PMID 31082164
- See also: Burn out an occupational phenomen — https://www.who.int/news/item/28-05-2019-burn-out-an-occupational-phenomenon-international-classification-of-diseases